CLINICAL TRIAL: NCT01911299
Title: Choline Supplementation in Children With Fetal Alcohol Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jennifer Thomas, Associate Director - Center for Behavioral Teratology, San Diego State University, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBT-choline-1
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Fetal Alcohol Spectrum Disorders; Fetal Alcohol Syndrome; Partial Fetal Alcohol Syndrome; Alcohol-related Neurodevelopmental Disorder; Prenatal Alcohol Exposure
Keywords: Choline; Glycerophosphocholine; Choline alphoscerate; Fetal alcohol spectrum disorders; Fetal alcohol syndrome; Partial fetal alcohol syndrome; Alcohol-related neurodevelopmental disorder; Prenatal alcohol exposure; Fetal Alcohol Effects; Pregnancy Complications; Alcohol-Induced Disorders; Alcohol-Related Disorders; Central Nervous System Agents; Therapeutic Uses
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Pregnancy Complications; Alcohol-Induced Disorders; Alcohol-Related Disorders | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Choline (Experimental): Liquid glycerophosphocholine (GPC) supplement
  Interventions: Dietary Supplement: Choline
- Placebo (Placebo Comparator): Liquid placebo supplement
  Interventions: Dietary Supplement: placebo supplementation consisting of vegetable glycerin (50% by volume) and deionized water

INTERVENTIONS:
Dietary Supplement: Choline — 5.25 ml of liquid glycerophosphocholine (approximately 1240 mg GPC), equivalent to 625 mg of choline
  Arms: Choline
Dietary Supplement: placebo supplementation consisting of vegetable glycerin (50% by volume) and deionized water
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether choline supplementation can improve cognitive functioning of children with prenatal alcohol exposure.

DETAILED DESCRIPTION:
Despite the known damaging effects of alcohol on the developing fetus and the presence of warning labels on alcoholic beverages, many pregnant women continue to drink alcohol. The consequences include a range of physical, neurological, and behavioral effects referred to as fetal alcohol spectrum disorders (FASD). Unfortunately, there are currently no comprehensive treatments for individuals with FASD. This pilot study will examine whether a nutritional intervention could reduce the severity of cognitive deficits associated with prenatal alcohol exposure. Choline is an essential nutrient, necessary for brain and behavioral development. Animal studies have shown that prenatal or early postnatal choline supplementation can lead to long-lasting cognitive enhancement. Similarly, choline supplementation improves cognitive outcomes among rats exposed to alcohol during development, even when administered postnatally and after alcohol exposure has occurred. The present experiment translates these findings to a clinical population of individuals exposed to heavy prenatal alcohol exposure. Subjects will be randomly assigned to receive daily choline supplementation or placebo control for a period of 6 weeks (approximately 20 subjects per group). Performance on neuropsychological tasks that measure cognitive functioning will be measured prior to treatment and at 6 weeks. These data will provide important information regarding a potential nutritional intervention for fetal alcohol spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histories of prenatal alcohol exposure (by review of medical, legal, or social service records or maternal report, if available; information about levels and timing of exposure will be inquired, but not necessary for inclusion)
* English as primary language

Exclusion Criteria:

* Significant physical (e.g., uncorrected visual impairment, hemiparesis) or psychiatric (e.g., psychosis) disability that would prohibit participation
* History of neurological condition (e.g., epilepsy)

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive function as measured by performance on neuropsychological tasks of learning/memory, executive functions, and attention | Baseline and 6 weeks

SECONDARY OUTCOMES:
Children's Behavior Checklist (CBCL), Behavioral Rating Inventory of Executive Function (BRIEF) | Baseline and 6 weeks
  Parent questionnaires about children's behavioral functioning will assess any behavioral changes over the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D. Thomas, Ph.D., Principal Investigator — San Diego State University
Locations (1):
- Center for Behavioral Teratology, San Diego State University, San Diego, California, United States

REFERENCES:
- [Derived] Nguyen TT, Risbud RD, Mattson SN, Chambers CD, Thomas JD. Randomized, double-blind, placebo-controlled clinical trial of choline supplementation in school-aged children with fetal alcohol spectrum disorders. Am J Clin Nutr. 2016 Dec;104(6):1683-1692. doi: 10.3945/ajcn.116.142075. Epub 2016 Nov 2. PMID 27806977